CLINICAL TRIAL: NCT02913469
Title: The Effects of Morphine on Loading-dose Ticagrelor in Patients With ST-segment Elevation Myocardial Infarction Before Primary Percutaneous Coronary Interven Tion
Brief Title: Effects of Morphine on Loading-dose Ticagrelor in Patients With ST-segment Elevation Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Morphine & Ticagrelor
Record Dates: First submitted 2016-09-09; First posted 2016-09-23 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: Morphine，Ticagrelor，STEMI，PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Morphine; Metoclopramide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- morphine+metoclopramide (Experimental): administrated intravenous morphine 5mg and metoclopramide 10mg
  Interventions: Drug: Morphine; Drug: metoclopramide
- morphine (Active Comparator): avenous morphine 5mg and 0.9%normal saline 2ml
  Interventions: Drug: Morphine; Drug: saline
- metoclopramide (Sham Comparator): intravenous metoclopramide 10mg and 0.9%normal saline 2ml
  Interventions: Drug: metoclopramide; Drug: saline
- placebo (Placebo Comparator): intravenous 0.9%normal saline 2mland 0.9%normal saline 2ml
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Morphine — The patients in group A would be administrated intravenous morphine 5mg
  Other Names: morphine hydrochloride
  Arms: morphine; morphine+metoclopramide
Drug: metoclopramide — the patients in group C would be administrated intravenous metoclopramide 10mg
  Other Names: Pasprtin
  Arms: metoclopramide; morphine+metoclopramide
Drug: saline — the patients in group D would be administrated intravenous 0.9%normal saline 2mland 0.9%normal saline 2ml.
  Other Names: Physiological Saline
  Arms: metoclopramide; morphine; placebo

SUMMARY:
Percutaneous coronary intervention(PCI) has become the first choice for STEMI patients.According to the current guidelines,dual antiplatelet therapy with a P2Y12 receptor inhibitor and aspirin ,and intravenous injection of morphine therapy for chest pain relief in necessity play a pivotal role in the treatment of patients with ST elevation myocardial infarction before primary percutaneous coronary intervention.And ticagrelor is recommended in patients with ST segment elevation myocardial infarction undergoing PCI, with class IB indication.Therefore coadministration of morphine and ticagrelor are commonplace.Currently, some studies have found that morphine delayed and attenuated exposure to ticagrelor,but it is not clear of the pathogenesis of it.Some researchers say that morphine results in a weaker and retarded antiplatelet effect of ticagrelor in STEMI patients before PCI by inhibition of gastrointestinal peristalsis and causing vomiting.The study is aimed at exploring whether morphine delay and attenuate exposure to ticagrelor and its antiplatelet effect.In addition, the trial will explore the possible mechanism which morphne delay and attenuate exposure to ticagrelor in patients with ST-segment elevation myocardial infarction before PCI.

DETAILED DESCRIPTION:
The study is a single center, randomized, single-blind, controlled trial.From September 1st, 2014 to February 10, 2016，patients with STEMI who prepared to accept PCI were screened according to the inclusion criteria. All patients for eligibility for the study received orally a 300 mg loading dose (LD) of plain aspirin and a 180mg loading dose (LD) of plain ticagrelor and then signed a written informed consent to participate in the study.Then,the patients were randomly assigned to four treatment groups.The patients in group A would be administrated intravenous morphine 5mg and metoclopramide 10mg,the patients in group B would be administrated intravenous morphine 5mg and 0.9%normal saline 2ml,the patients in group C would be administrated intravenous metoclopramide 10mg and 0.9%normal saline 2ml, the patients in group D would be administrated intravenous 0.9%normal saline 2mland 0.9%normal saline 2ml. Subsequently，all patients would received orally plain aspirin 100mg once a day and plain ticagrelor 90mg twice a day and 1 month of follow-up.The investigators would calculate the platelet response index before LD and 0.5h,2h,8h after LD by platelet vasodilator-stimulated phosphoprotein phosphorylation assay with flow cytometry instrument(BD FACS Calibur). The primary study end-point was platelet response index by PRI VASP 2 hours after LD. Secondary end-points were (1) The platelet response index by PRI VASP half an hour and 8 hours after LD.(2)Record the electrocardiogram changes(the incidence of a 70% reduction after PCI ,TIMI flow of crime vessels(TIMI flow frames),the incidence of acute/subacute thrombotic events,the incidence of major adverse cardiovascular and cerebrovascular events,the incidence of primary and secondary bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedures
2. Male or female aged from 18 to 80 years old
3. Patients with STEMI scheduled to undergo PCI.

Exclusion Criteria:

1. Hypersensitivity to the active substance or to any of the excipients
2. Active bleeding or bleeding diathesis
3. Previous transient ischemic attack
4. Antiplatelet (clopidogrel, prasugrel, ticagrelor) administration in the week before the index event
5. Known relevant hematological conditions
6. Left ventricular ejection fraction ≤ 30%
7. Renal failure with creatinine ≥ 3 mg/dl
8. History of liver disease
9. Increased risk of bradycardia
10. Concomitant therapy with drugs known to interfere with CYP3A4 metabolism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2014-12-12 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Platelet Reactivity Index(PRI) Measured by VASP-P | 2 hours after the loading dose of ticagrelor
  Vasodilator-stimulated phosphoprotein(VASP) phosphorylation, a measure of P2Y12 receptor reactivity, was determined by flow cytometry with the use of the Platelet VASP-FCM Kit (Stago, France)and recorded as the platelet reactivity index

SECONDARY OUTCOMES:
Platelet Reactivity Index (PRI) Measured by VASP-P | 0.5hour,8hours after the loading dose of ticagrelor
the incidence of major adverse cardiovascular and cerebrovascular events | follow-up for 30 days after the loading dose of ticagrelor

CONTACTS AND LOCATIONS:
Overall Officials: huiliang liu, MD, Study Chair — CHINESE ARMED POLICE FORCE GENRAL HOSPITAL
Locations (1):
- Cardiology Department, Chinese Armed Police Force Genral Hospital, Beijing China, Beijing, China

IPD SHARING:
Plan to Share IPD: No